CLINICAL TRIAL: NCT01191619
Title: Comparison of Two Insertion Techniques of Proseal Laryngeal Mask Airway by Unskilled Personnel in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Seoul National University Bundang Hospital, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: B1006/104-004
Record Dates: First submitted 2010-08-05; First posted 2010-08-31 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-07

CONDITIONS: Airway Management
Keywords: McIvor retractor; Proseal laryngeal mask airway

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- McIvor group (Experimental): groups in which proseal laryngeal mask airway is inserted with McIvor retractor.
  Interventions: Procedure: McIvor retractor

INTERVENTIONS:
Procedure: McIvor retractor — The Mclvor blade- guided technique (McIvor group) involved the following steps. The PLMA was lubricated on the posterior aspect of the deflated mask with a water-based lubricant. The McIvor blade was fully inserted beneath the tongue of the patients. The tongue was lifted gently with the McIvor blade and PLMA was introduced into a space between the McIvor blade and maxillary incisors holding the bite block of the PLMA. The PLMA was advanced into the hypopharynx until definite resistance was felt and McIvor blade was removed.
  Other Names: McIvor group

SUMMARY:
The ProSeal laryngeal mask airway (PLMA) is one of the alternative methods for effective airway management. It is an advanced form of laryngeal mask airway(LMA) with a softer and larger cuff to improve sealing and a drain tube to permit venting of the stomach. However, the larger cuff is more difficult to save space for insertion in the mouth and is more likely to fold over. Particularly, a relatively large tongue, a floppy epiglottis, a cephalad and more anterior larynx and frequent presence of tonsillar hypertrophy may disturb PLMA insertion in pediatric patients. The manufacturer recommends inserting PLMA using digital manipulation or with an introducer, but these techniques have lower success rates compared to those of LMA insertion.

McIvor blade is a tongue retractor with a thin and curved blade and a flat handle. It is used to secure the operating field by pressing tongue during tonsillectomy. The investigators hypothesized that McIvor blade would provide more space in the mouth for PLMA insertion, and therefore it could improve the PLMA insertion as well as reducing injuries to the pharyngeal wall. The investigators compared the success rate and the incidence of complications of the digital technique with those of McIvor blade-guided insertion by unskilled anesthesia residents.

DETAILED DESCRIPTION:
Rapid and successful airway management is important for the patient's outcome in emergency care. Tracheal intubation with an endotracheal tube is the gold standard for airway management, but tracheal intubation by paramedical staff in pre-hospital setting can be time-consuming and difficult. The ProSealTM laryngeal mask airway (PLMA) is one of the alternative methods for effective airway management. It is an advanced form of laryngeal mask airway(LMA) with a softer and larger cuff to improve sealing and a drain tube to permit venting of the stomach. However, the larger cuff is more difficult to save space for insertion in the mouth and is more likely to fold over. Particularly, a relatively large tongue, a floppy epiglottis, a cephalad and more anterior larynx and frequent presence of tonsillar hypertrophy may disturb PLMA insertion in pediatric patients. The manufacturer recommends inserting PLMA using digital manipulation or with an introducer, but these techniques have lower success rates compared to those of LMA insertion. The first attempt success rate of PLMA insertion by inexperienced personnel was reported to be 83%. Several techniques have been introduced to improve the insertion success rate; the use of fiberoscopy, gum-elastic bougie, and a suction catheter. However, all of them can not save enough oral space for PLMA insertion and it would not be easy for the unskilled personnel to use them in emergency situations. A larger space between tongue and retropharynx, not being accompanied with an index finger for insertion would make make it easier for the unskilled personnel to insert the PLMA.

McIvor blade is a tongue retractor with a thin and curved blade and a flat handle. It is used to secure the operating field by pressing tongue during tonsillectomy. We hypothesized that McIvor blade would provide more space in the mouth for PLMA insertion, and therefore it could improve the PLMA insertion as well as reducing injuries to the pharyngeal wall. We compared the success rate and the incidence of complications of the digital technique with those of McIvor blade-guided insertion by unskilled anesthesia residents.

ELIGIBILITY:
Inclusion Criteria:

* healthy pediatric patients undergoing surgery under general anesthesia

Exclusion Criteria:

* pediatric patients with a known or predicted difficult airway, recent sore throat, mouth opening less than 2.5 cm, or at risk of aspiration

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
the success rate of proseal laryngeal mask airway (PLMA) insertion | at the time of insertion of PLMA
  immediately after the insertion of PLMA

SECONDARY OUTCOMES:
the incidence of complications following PLMA insertion | after the removal of PLMA, and 1 day after surgery
  blood staining: after the removal of PLMA; sore throat: 1 day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Hwang, MD, Principal Investigator — Fellow
Locations (1):
- Seoul National University Bundang Hospital, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Hwang J, Han S, Hwang J, Oh A, Park S, Kim J. The McIvor blade improves insertion of the LMA ProSeal in children. Can J Anaesth. 2011 Sep;58(9):796-801. doi: 10.1007/s12630-011-9540-4. Epub 2011 Jun 21. PMID 21691935